CLINICAL TRIAL: NCT03255759
Title: Assessment of the Use and Impact of a Molecular Identification Assay in the Diagnosis and Management of Bloodstream Infections at in Healthcare Settings in Princess Marina Hospital, Botswana
Brief Title: Actionable Results: Bloodstream Infection Molecular Assay Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08821/1/1
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Bloodstream Infection
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Molecular dx arm (Active Comparator): Positive blood cultures are tested using a molecular ID system in addition to the standard of care (biochemical identification)
  Interventions: Diagnostic Test: Multiplex molecular diagnostic assay
- Standard of care arm (No Intervention): Positive blood cultures are treated as per normal lab protocol (biochemical identification)

INTERVENTIONS:
Diagnostic Test: Multiplex molecular diagnostic assay — To assess the added value and acceptability of a multiplexed molecular diagnostic assay in the identification of pathogens in patients presenting with bacteremia at hospitals in LMICs, and to assess health care providers' satisfaction with the assay.
  Arms: Molecular dx arm

SUMMARY:
A number of rapid panel-based molecular assays for direct organism identification and resistance characterization in positive blood culture bottles are now commercially available. They have been shown to improve accuracy and decrease the time-to-result, allowing targeted treatment in hospitalized patients with bacteraemia, in high-income countries (HICs). However, these molecular assays are add-on tests performed in addition to conventional testing, increasing the complexity of diagnostic algorithms and costs of patient care. Conventional organism identification includes performing a Gram stain, biochemical identification and phenotypic drug susceptibility testing. The FilmArray Blood Culture Identification (BioFire, USA) is an example of a rapid panel-based molecular assay that combines nesting and multiplexing of PCR (nested multiplex PCR) to detect multiple pathogens simultaneously. There are limited data on how such tests impact patient management, health care costs and how they can better be incorporated into diagnostic algorithms.

The aim of this study is to assess the added value and acceptability of a multiplexed molecular diagnostic assay in the identification of pathogens in patients presenting with bacteremia at hospitals in LMICs, and to assess health care providers' satisfaction with the assay.

DETAILED DESCRIPTION:
The study will address the following questions:

1. What impact can we project if additional diagnostic information were to be provided to clinicians in terms of patient outcomes, costs, and antibiotic use?
2. What are the workflow constraints on returning diagnostic results to clinicians and/or antibiotic stewardship programs? Overall, the aim is to assess the added value and acceptability of a multiplexed molecular diagnostic assay in the identification of pathogens in patients presenting with bacteremia at hospitals in LMICs and to assess health care providers' satisfaction with the assay.

ELIGIBILITY:
Inclusion Criteria:

* For patients of Princess Marina Hospital: all participants who have a blood culture done as part of routine clinical care that is found to be positive through routine laboratory testing from Monday-Friday 8am-3pm (excluding holidays) will be eligible for inclusion in the study, regardless of age and co-morbidities.
* For the professionals making use of molecular testing: Attending physicians (paediatricians, internists, and physician trainees [residents, medical officers, interns]) caring for adults and children who are enrolled in the study, Microbiologists and microbiology technologists who have experience operating the BioFire FilmArray and/or traditional blood culture incubation systems at the laboratory.

Exclusion Criteria:

* For patients of Princess Marina Hospital: Individuals who have previously participated in the study by having a blood culture positive in the week prior will not be eligible to participate again within the 7-day time frame.
* For professionals making use of molecular testing: Individuals working with patients or laboratory samples at Princess Marina Hospital for less than one month will not be asked to participate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Time from blood collection to definitive treatment initiation (optimal treatment defined as time from blood culture collection to the initiation of a predetermined pathogen-specific antimicrobial therapy) | 1year
  The judgment as to whether antimicrobial treatment was effective or optimal will be assessed by two members of the study team (infectious disease specialists and/or microbiologists) blinded to treatment group. A third, blinded, party member will be available to adjudicate unresolved disagreements. The Principal Investigators will not be involved in outcome classification.

SECONDARY OUTCOMES:
Time from blood collection to initiation of effective antimicrobial therapy (initiation of antimicrobials active against the identified causative pathogen) | 1year
  The aim is to understand the reduction in time it takes clinical staff to act upon the result. Faster treatment is associated with reduced mortality.
Time from blood collection to pathogen identification | 1year
  The hypothesis is that faster identification will lead to faster action.
Proportion of patients with a confirmed diagnosis of bloodstream infection who are started on optimal antimicrobial therapy in the intervention compared to control arm. | 1year
  This outcome will inform how the inclusion of a faster diagnosis can support antibiotic stewardship efforts.
Frequency of discrepant results between molecular identification vs standard of care. | 1year
  Current panels are design for common pathogens in the USA and Europe and given that this is the first evaluation in Africa it will advice on the suitability.
Clinicians' satisfaction with the assay, predominantly in terms of time-to-result and actionable results. | 2month
  To inform future projects and help guide implementation efforts.
Laboratory professional satisfaction with the assay, predominantly in terms of ease of use and workflow. | 2month
  To inform future projects and help guide implementation efforts.
In-hospital mortality. | 1year
  Faster treatment is associated with reduced mortaltity and as a secondary outcome we want to assess the difference between standard of care and diagnostic intervention.
30-day mortality. | 1year
  Faster treatment is associated with reduced mortaltity and as a secondary outcome we want to assess the difference between standard of care and diagnostic intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pernica, MD, FRCPC, Principal Investigator — McMaster University; David Goldfarb, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana